CLINICAL TRIAL: NCT04634110
Title: Brigatinib Before Brain Irradiation Trial (B3i Trial): A Phase II Trial of Brigatinib Alone for Brain Metastases From ALK+ Lung Cancer
Brief Title: Brigatinib Before Brain Irradiation Trial (B3i Trial)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-2862.cc; P30CA046934 (NIH)
Record Dates: First submitted 2020-10-23; First posted 2020-11-18 (Actual); Results first posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-09

CONDITIONS: Brain Metastases; Lung Cancer
MeSH Terms: conditions — Brain Neoplasms; Lung Neoplasms | interventions — brigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients with ALK+ NSCLC and brain metastases (Experimental): Including patients with brain metastases from ALK (anaplastic lymphoma kinase) positive NSCLC (non-small cell lung cancer), who are either neurologically asymptomatic or who have only mild neurologic symptoms (RTOG [Radiation therapy Oncology Group] acute neurologic morbidity score 0-2) from their brain metastases, who are TKI (tyrosine kinase inhibitor) naïve or who have had prior exposure to crizotinib, but who are naïve to brigatinib and other ALK TKIs including alectinib, lorlatinib, and ceritinib.
  Interventions: Drug: Brigatinib

INTERVENTIONS:
Drug: Brigatinib — At day 1, all patients will be started on brigatinib 90 mg daily for 7 days, before escalating to 180 mg daily thereafter as tolerated.

SUMMARY:
This is a single arm phase II study of brigatinib alone for patients with brain metastases from anaplastic lymphoma kinase (ALK) positive non-small cell lung cancer (NSCLC), who have either not been treated previously with a tyrosine kinase inhibitor (TKI) targeting ALK or who have had prior exposure to crizotinib.

DETAILED DESCRIPTION:
In this single-arm phase II trial, patients with brain metastases from ALK+ NSCLC will be treated with brigatinib alone without upfront brain irradiation. Patients will have close monitoring with clinical follow up visits and brain magnetic resonance imaging (MRI) surveillance, which will maximize safety and allow for early treatment if disease progression is observed. If brigatinib alone can demonstrate high rates of CNS disease control, these data could support a strategy of upfront brigatinib alone for carefully selected patients with brain metastases from ALK+ NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form.
2. Stated willingness to comply with all study procedures and be available for the duration of the study.
3. Ability to take and retain oral medications.
4. Age ≥18 years.
5. Patients with ALK+ lung cancer with evidence of ≥1 previously untreated brain metastases on brain MRI. Prior therapy (radiation or surgery) for brain metastases is allowed. However, patients must have ≥1 previously untreated at the time of enrollment.
6. Patients may be ALK TKI naïve OR have had prior crizotinib therapy.
7. Patients may be included if they are asymptomatic from their brain metastases (RTOG/EORTC grade 0) or if they have mild symptoms from their brain metastases not to exceed RTOG/ EORTC grade 1 or 2 (Grade 1: Fully functional status (i.e. able to work) with minor neurological findings, no medication needed; Grade 2: Neurological findings present sufficient to require home care / nursing assistance may be required / medications including steroids/anti-seizure agents may be required) (Cox, James D., et al "Toxicity criteria of the radiation therapy oncology group (RTOG) and the European organization for research and treatment of cancer (EORTC)." International Journal of Radiation Oncology• Biology• Physics 31.5 (1995): 1341-1346).
8. Neurologically symptomatic patients must not require immediate surgical or radiation therapy for their symptoms, as decided by an investigator.
9. Have an Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
10. Have adequate organ function, as determined by

    * ALT/AST ≤2.5 × upper limit of normal (ULN); ≤5 × ULN is acceptable if liver metastases are present
    * Total serum bilirubin ≤1.5 × ULN (<3.0×ULN for patients with Gilbert syndrome)
    * Estimated glomerular filtration rate (eGFR) ≥30 mL/min/1.73 m2, using the modification of diet in renal disease (MDRD) equation
    * Serum lipase/amylase ≤1.5 × ULN
    * Absolute neutrophil count (ANC) ≥1.5 × 109/L
    * Platelet count ≥75 × 109/L
    * Hemoglobin ≥9 g/dL
11. For females of childbearing potential, have a negative pregnancy test documented prior to initiating brigatinib.
12. For female and male patients who are fertile, agree to use 2 effective methods of contraception with their sexual partners from the time of signing the informed consent through 4 months after the last dose of study drug, or agree to completely abstain from heterosexual intercourse. Brigatinib may decrease effectiveness of hormonal contraceptives, therefore, women are recommended to use non-hormonal methods of contraception. Highly effective non-hormonal birth control for women of child bearing potential with male partners includes:

    * Sexual abstinence (no sexual intercourse)
    * Intrauterine device (IUD) or intrauterine system (IUS)
    * Bilateral tubal ligation (both tubes tied)
    * Vasectomized partner
13. Male patients, even if surgically sterilized (i.e., status post-vasectomy) must agree to 1 of the following:

    * Practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug, or completely abstain from heterosexual intercourse.

Exclusion Criteria:

1. Patients who have received prior brigatinib therapy or other CNS-penetrant ALK TKIs, including alectinib, lorlatinib, or ceritinib.
2. RTOG/EORTC Acute CNS symptoms, grade 3 and 4 (Grade 3: Neurological findings requiring hospitalization for initial management; Grade 4: Serious neurological impairment that includes paralysis, coma, or seizures > 3 per week despite medication / hospitalization required).
3. Currently pregnant, planning a pregnancy during the study period, or breastfeeding.
4. Have clinically significant, uncontrolled cardiovascular disease per investigator, specifically including, but not restricted to:

   1. Myocardial infarction (MI) within 6 months prior to the first dose of study drug
   2. Unstable angina within 6 months prior to first dose of study drug
   3. Clinically significant congestive heart failure (CHF) within 6 months prior to first dose of study drug
   4. History of clinically significant atrial or ventricular arrhythmia (including clinically significant bradyarrhythmia), as determined by the treating physician
   5. Cerebrovascular accident or transient ischemic attack within 6 months prior to first dose of study drug
5. Have uncontrolled hypertension per the investigator. Patients with persistent hypertension of systolic ≥140 or diastolic ≥90 mm Hg should be under treatment on study entry to control blood pressure.
6. Have a history or the presence at baseline of pulmonary interstitial disease, drug-related pneumonitis, or radiation pneumonitis.
7. Have an ongoing or active infection, including, but not limited to, the requirement for intravenous (IV) antibiotics.
8. Have a known history of human immunodeficiency virus (HIV) infection. Testing is not required in the absence of history.
9. Have a known or suspected hypersensitivity to brigatinib or its excipients.
10. Additional systemic therapies for the treatment of lung cancer may not be taken concomitantly with brigatinib (eg, TKIs, immunotherapy, chemotherapy). No washout period is required for prior therapy.
11. Have malabsorption syndrome or other GI illness that could affect oral absorption of brigatinib.
12. Have any condition or illness that, in the opinion of the investigator, would compromise patient safety or interfere with the evaluation of brigatinib.
13. Received systemic treatment with strong cytochrome p-450 (cyp)3a inhibitors, strong cyp3a inducers, or moderate cyp3a inducers within 14 days before enrollment.
14. Had major surgery within 30 days of the first dose of brigatinib. Minor surgical procedures such as catheter placement or minimally invasive biopsies are allowed.
15. Have been diagnosed with another primary malignancy other than NSCLC, except for adequately treated nonmelanoma skin cancer or cervical cancer in situ; definitively treated nonmetastatic prostate cancer; or patients with another primary malignancy who are definitively relapse-free with at least 3 years elapsed since the diagnosis of the other primary malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chad Rusthoven, MD, Principal Investigator — University of Colorado, Denver
Locations (3):
- United States (3):
  - City of Hope, Duarte, California
  - University of Colorado Hospital, Aurora, Colorado
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With ALK+ NSCLC and Brain Metastases
Started | 1
Completed (Subject did not complete treatment) | 0
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Patients With ALK+ NSCLC and Brain Metastases
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 57 [57 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Meet Disease Control Rate (DCR) Criteria of Brain Metastases at 3 Months
Description: DCR is defined as complete response (CR), partial response (PR), or stable disease (SD) as defined by the RANO-BM (Response Assessment in Neuro-Oncology Criteria - Brain Metastases) criteria.
Time Frame: 13-week MRI ±7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With ALK+ NSCLC and Brain Metastases
Number analyzed (Participants) | 1
Participants | 1

2. Secondary Outcome: Time Until Progression With Brigatinib Alone (Part 1)
Description: Time until any CNS progressive disease (PD) by RANO-BM criteria and rates at follow up intervals
Time Frame: up to 24 months
Population: Trial was terminated early due to low accrual. No data were collected for this outcome measure because the patient was only followed for 13 weeks, and progression did not occur during this time.
Arm/Group | Patients With ALK+ NSCLC and Brain Metastases
Number analyzed (Participants) | 0

3. Secondary Outcome: Time Until Progression With Brigatinib Alone (Part 2)
Description: Time until any local PD (i.e., in brain lesions identified at the time of enrollment) by RANO-BM criteria and rates at follow up intervals
Time Frame: up to 24 months
Population: as for outcome 2
Arm/Group | Patients With ALK+ NSCLC and Brain Metastases
Number analyzed (Participants) | 0

4. Secondary Outcome: Time Until Progression With Brigatinib Alone (Part 3)
Description: Time until any distant brain PD (i.e., new brain lesions that were not present at the time of enrollment) by RANO-BM criteria and rates at follow up intervals
Time Frame: up to 24 months
Population: as for outcome 2
Arm/Group | Patients With ALK+ NSCLC and Brain Metastases
Number analyzed (Participants) | 0

5. Secondary Outcome: Time Until Progression With Brigatinib Alone (Part 4)
Description: Time until progression at any site using RANO-BM for intracranial disease and RECIST for extracranial disease and rates at follow up intervals
Time Frame: up to 24 months
Population: as for outcome 2
Arm/Group | Patients With ALK+ NSCLC and Brain Metastases
Number analyzed (Participants) | 0

6. Secondary Outcome: Overall Survival With a Strategy of Brigatinib Alone
Description: Time until death from any cause and rates at follow up intervals
Time Frame: up to 24 months
Population: Trial was terminated early due to low accrual. No data were collected for this outcome measure because the patient was only followed for 13 weeks and did not die.
Arm/Group | Patients With ALK+ NSCLC and Brain Metastases
Number analyzed (Participants) | 0

7. Secondary Outcome: Time Until Brain Metastases-Specific Mortality
Description: Defined as time to intracranial progression as a component of cause of death and rates at follow up intervals
Time Frame: up to 24 months
Population: Trial was terminated early due to low accrual. No data were collected for this outcome measure because the patient was only followed for 13 weeks, and neither progression nor death occurred during this time.
Arm/Group | Patients With ALK+ NSCLC and Brain Metastases
Number analyzed (Participants) | 0

8. Secondary Outcome: Brain Metastases Objective Response Rates (ORR) With Brigatinib Alone
Description: Cumulative rate of best responses individually for complete response (CR), partial response (PR), stable disease (SD), by RANO-BM criteria
Time Frame: up to 24 months
Population: Trial was terminated early due to low accrual. No data were collected for this outcome measure because the patient was only followed for 13 weeks.
Arm/Group | Patients With ALK+ NSCLC and Brain Metastases
Number analyzed (Participants) | 0

9. Secondary Outcome: Time Until the Administration of WBRT With Brigatinib Alone
Description: Time until the administration of whole brain-radiotherapy (WBRT) and rates at follow up intervals
Time Frame: up to 24 months
Population: Trial was terminated early due to low accrual. No data were collected for this outcome measure because the patient was only followed for 13 weeks and did not receive WBRT before trial termination.
Arm/Group | Patients With ALK+ NSCLC and Brain Metastases
Number analyzed (Participants) | 0

10. Secondary Outcome: Longitudinal Changes in Quality of Life With Brigatinib Alone
Description: Quality of life will be assessed using standardized QOL metrics (EORTC QLQ C30/BN 20)
Time Frame: up to 24 months
Population: Trial was terminated early due to low accrual. No scores were computed for this outcome measure because the patient was only followed for 13 weeks out of the intended 104 weeks and longitudinal changes could not be analyzed.
Arm/Group | Patients With ALK+ NSCLC and Brain Metastases
Number analyzed (Participants) | 0

11. Other Pre Specified Outcome: Analysis of Blood at Baseline and at Progression to Correlate With Clinical Outcomes
Description: Evaluation of cfDNA at baseline and progression to correlate with clinical outcomes, including incidence of disease recurrence per RANO-BM and RECIST 1.1, survival status by percentage of patients alive at 2 years, and patient rating of quality of life per EORTC QLQ-BN20 and EORTC QLQ-C30 questionnaires.
Time Frame: up to 24 months
Population: Trial was terminated early due to low accrual. No data were collected for this outcome measure because the patient was only followed for 13 weeks, and no progression occurred during this time.
Arm/Group | Patients With ALK+ NSCLC and Brain Metastases
Number analyzed (Participants) | 0

12. Other Pre Specified Outcome: Characterization of Corticosteroid Administration Before and After Brigatinib Initiation
Description: Quantification of the agent and dosage of corticosteroids at each study assessment
Time Frame: up to 24 months
Population: Trial was terminated early due to low accrual. No data were collected for this outcome measure because the patient was only followed for 13 weeks and had not been administered any corticosteroids during this time.
Arm/Group | Patients With ALK+ NSCLC and Brain Metastases
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 13 weeks
Arm/Group | Patients With ALK+ NSCLC and Brain Metastases
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With ALK+ NSCLC and Brain Metastases (N=1)
Non-Cardiac Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (3)
Somnolence (General disorders) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Hyponatremia (Blood and lymphatic system disorders) | 1 (1)
CPK increased (Blood and lymphatic system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Vocal Cord Paralysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
xerosis (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
1 subject enrolled then study terminated due to low accrual. No further analyses completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-29): https://cdn.clinicaltrials.gov/large-docs/10/NCT04634110/Prot_SAP_000.pdf